CLINICAL TRIAL: NCT05832424
Title: Feasibility and Acceptability of a Telehealth Intervention Among Women With Perinatal Depression/Anxiety and Substance Use Risk.
Brief Title: Feasibility and Acceptability of a Telehealth Intervention Among Women With Perinatal Mental Health
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boise State University (Other)
Responsible Party: Principal Investigator, Ryoko Kausler, Assistant Professor, Boise State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: bsu0307
Record Dates: First submitted 2023-03-07; First posted 2023-04-27 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Perinatal Depression; Perinatal Anxiety; Substance Use; Telehealth
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- UPLIFT Telehealth Intervention (Experimental): The telehealth group intervention will be delivered using Zoom. Participants will attend facilitated weekly, 1-hour sessions for 8 weeks. The sessions follow a standardized, manualized program based on cognitive-behavioral therapy (CBT) and mindfulness-based practice (MBP)-therapies widely accepted and used by mental health providers for the treatment and prevention of depression and substance use. The study team have tailored this intervention for use in a pregnant population.
  Interventions: Behavioral: UPLIFT program

INTERVENTIONS:
Behavioral: UPLIFT program — The telehealth group intervention will be delivered using Zoom. Participants will attend facilitated weekly, 1-hour sessions for 8 weeks. The sessions follow a standardized, manualized program based on cognitive-behavioral therapy (CBT) and mindfulness-based practice (MBP)-therapies widely accepted and used by mental health providers for the treatment and prevention of depression and substance use. The study team have tailored this intervention for use in a pregnant population.

SUMMARY:
The goal of this pilot feasibility/acceptability study is to evaluate the effectiveness of a telehealth approach to increase access to services and reduce depression/anxiety symptoms and risk of substance use in a population of women with perinatal depression/anxiety and elevated substance use risk. The main questions it aims to answer are:

* Assess the acceptability and feasibility of a telehealth approach to deliver an 8-week evidence-based group intervention to women with perinatal depression/anxiety and mild to moderate substance use risk.
* Obtain preliminary data on treatment response to a telehealth 8-week evidence-based group intervention.

Participants will participate in an 8-week evidence-based group intervention and complete the study questionnaire including depression severity, treatment adherence, and substance use risk which will be evaluated at baseline, post-intervention, and 2-month follow-up.

DETAILED DESCRIPTION:
The prevalence of substance use during pregnancy is a population health concern, particularly with the increasing use of opioids and marijuana during pregnancy. At the same time, perinatal depression occurs in 12% to 15% of pregnant and postpartum women. Recent studies indicate that approximately 45% of women with perinatal depression/anxiety report substance use during pregnancy. Likewise, up to 65% of women with perinatal substance use screen positive for symptoms of perinatal depression/anxiety or have a history of depression/anxiety, suggesting that this population is at increased substance-use risk. It is critical to deliver treatment for perinatal mood disorders that also addresses substance-use risk. During the coronavirus disease (COVID-19) pandemic, data suggest a significant relationship between self-reported mental/emotional health, stress, and depressive symptoms and substance use among pregnant women due to intense emotional distress with feelings of uncertainty during the pandemic. Therefore, it is critical to deliver treatment for perinatal mood disorders that also addresses substance-use risk, which refers to current or previous substance use that does not rise to the level of a substance use disorder but does have a known association with progression to a diagnosis of substance use disorder. Effective nonpharmacological approaches (e.g., mindfulness based cognitive-behavioral therapy - MBCT) exist for perinatal depression/anxiety and substance use. However, studies typically evaluate these interventions for perinatal depression/anxiety and substance use separately. Furthermore, perinatal depression rates in rural areas are nearly double, but specialty care for perinatal depression/anxiety and/or substance-use risk are rarely available to childbearing women in rural communities. Although stigma towards perinatal substance use exists in both urban and rural settings, lack of anonymity in rural settings prevent to seek the care of substance use. It is imperative to increase access to mental health services for women in rural areas affected by perinatal depression/anxiety with substance-use risk.

Telehealth is an innovative approach to increase access to therapies such as MBCT for women with perinatal depression/anxiety and for those with increased substance-use risk. Women with perinatal depression/anxiety consider cost and treatment type when seeking care for perinatal depression/anxiety, thus it is important to identify cost-effective preventative care and types of treatment, especially nonpharmacological approaches for this population to increase access of care. The success in using a videoconferencing system to deliver a wide range of care suggests that there is high potential for telehealth to deliver effective and affordable mental health services to women, including in low-resource settings and rural communities. In addition, studies demonstrated the feasibility and acceptability of a group telehealth intervention to deliver MBCT to women experiencing perinatal depressive symptoms. However, there is little evidence indicating that a telehealth approach is acceptable or feasible in a population of women who also have elevated substance-use risk. This study is grounded in a conceptual framework for associations between vulnerability, response, health outcomes, and a technology acceptance model to predict the acceptability of the telehealth approach. A long-term goal of the proposed study is to evaluate the effectiveness of a telehealth approach to increase access to services, improve treatment adherence, and reduce substance use in a population of women with perinatal depression/anxiety and elevated substance use risk. The proposed study will enroll 30 women with known perinatal depression/anxiety symptoms and self-reported substance-use risk into a telehealth intervention group. The specific aims of the study are to:

Aim 1: Assess the acceptability and feasibility of a telehealth approach to deliver an 8-week evidence-based group intervention to women with perinatal depression/anxiety and mild to moderate substance-use risk. Methods: Pregnant and postpartum women (up to 1 year) who screen positive for mild to moderate symptoms of depression (score of 9-20 on the Edinburgh Postnatal Depression Scale - EPDS) and self-reported low to moderate substance use risk (NIDA Quick/Modified ASSIST scores 0-27) will be enrolled in an evidence-based intervention using a telehealth group videoconferencing platform. Women will continue with standard care while attending weekly 1-hour sessions. Feasibility and acceptability will be measured as follows: (1) the number of eligible women who agree to participate in the telehealth intervention, (2) the number of sessions attended, (3) time to and number of participant dropouts, and (4) direct feedback from participants about their experiences with the program (telehealth focus groups and individual surveys).

Aim 2: Obtain preliminary data on treatment response to a telehealth 8-week evidence-based group intervention. Methods: Measures of depression severity, treatment adherence, and substance use risk will be evaluated at baseline, post-intervention, and 2-month follow-up. Measures include the EPDS, General Anxiety Disorder (GAD) -7, and participant reports of substance use risk using a NIDA Quick/Modified ASSIST.

The proposed study will advance the field by establishing whether a telehealth intervention is feasible and acceptable to women with perinatal depression/anxiety and elevated substance-use risk in their communities. Also, this study aligns with programmatic priorities focused on substance abuse and mental health as well as assessing how COVID-19 affects a vulnerable population. Pregnancy can be a motivating time for a woman to seek treatment associated with perinatal depression/anxiety with substance-use risk, but access to effective specialty services is a frequent barrier. Telehealth holds promise for increasing access to mental health services and prevention of increased substance-use risk.

ELIGIBILITY:
Inclusion Criteria:

* Women 18 and older who, at the time of enrollment
* Have a viable pregnancy or who are up to 12 months postpartum,
* Read and understand English, and
* Have an access to electronic device with internet access.

And who have at least one of the following risk factors for perinatal depression/anxiety:

* Have an Edinburgh Postnatal Depression Scale (EPDS) score of 9-20,
* History of depression or anxiety,
* Have experienced two or more significant life events that put them at risk for developing depression (measured on the screening questionnaire),
* Have an NIDA Quick Screen and answered "yes" with any choices,
* Have a total score of NIDA Modified ASSIST 0-26 (mild to moderate risk) and report the use of common substances (cannabis, prescription opioids, inhalants, prescribed stimulants, and sedatives or sleeping pills) based on NIDA-Modified ASSIST.

Exclusion Criteria:

* Less than 18 years old
* Have an EPDS score > 20
* Have a NIDA Modified ASSIST score > 26;
* Have a current diagnosis of a serious mental illness, such as psychosis, schizophrenia, bipolar disorder, severe depression, or suicidality
* Have a current diagnosis of substance use disorder; or
* Currently use street opioids, cocaine, methamphetamine, and/or hallucinogens based on NIDA-Modified ASSIST

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-03-15 (Estimated); Primary Completion 2025-01-22 (Estimated); Study Completion 2025-01-22 (Estimated)

PRIMARY OUTCOMES:
Feasibility of Telehealth - Enrollment Number | Recruitment
  The investigators will measure feasibility by the number of participants who agree to participate in the study. The proposed study will provide point estimates and confidence intervals (CIs) for use in a larger, fully powered trial. The recruitment rate will inform population point estimates and 95% CIs for sample measures. For example, with an estimate of 50% recruitment rate (60 assessed), this provides a point of estimate of 50% with a CI of +/- 13%.
Feasibility of Telehealth - Number of Sessions Attended | During 8-weeks intervention
  The investigator will measure feasibility by the number of sessions attended by participants. Attendance will be collected via REDCap to see out of 8 lessons, how many lessons participants attended.
Feasibility of Telehealth - Drop out rate | Through study completion, an average of 4 months
  The investigator will measure feasibility by the dropout rate. When the participant decides to drop out, the investigators will mark the participant as "dropped" and calculate drop out rate by the number of participants who "dropped" during the study time divided by the number of participants enrolled.
Feasibility of Telehealth - Drop out pattern | Through study completion, an average of 4 months
  The investigator will measure feasibility by the dropout patterns. When the participant decides to drop out, the investigator will ask for the reason and collect the information if the participant chooses to disclose it.
Acceptability of Telehealth- Satisfaction/Feedback | After completion of the intervention (8-weeks)
  The investigator will measure acceptability by utilizing satisfaction/feedback surveys administered at the study exit regardless of whether the individual has completed the intervention. Both ranked, and open-ended responses will assess satisfaction with the intervention overall; satisfaction with the videoconference system and group sessions; and feedback on usability and barriers to participation.
Acceptability of Telehealth- Focus group | Around 2 months post intervention (focus group)
  The investigator will measure acceptability by focus group interviews with 6 to 8 other participants, using Zoom. The purpose of the focus group is to collect data directly from participants regarding satisfaction with the program.

SECONDARY OUTCOMES:
Preliminary data on treatment response- Edinburgh Postnatal Depression Scale (EPDS) | pre intervention(after the informed consent), post intervention (at the end of intervention average 8 weeks after the intervention starts), 2 months post-intervention
  The Edinburgh Postnatal Depression Scale (EPDS) is a widely-used instrument for measuring depressive symptoms during both postpartum and pregnancy. The EPDS is an effective measure of depression in diverse populations of pregnant women. The range of scores is 0 to 30, where <9 indicates little to no depressive symptoms, 9-13 indicates increasing depressive symptoms, a score >13 indicates a positive screen for depression risk, and a score >20 indicates a high probability of a severe major depressive disorder.
Preliminary data on treatment response- General Anxiety Disorder (GAD)-7 | pre intervention(after the informed consent), post intervention (at the end of intervention average 8 weeks after the intervention starts), 2 months post-intervention
  The GAD-7 is a widely used, 7-item instrument considered to be a clinically meaningful measure for Generalized Anxiety Disorder (GAD).The range of scores is 0-21, with scores of 5, 10, and 15 taken as the cutoff points for, respectively, mild, moderate, and severe anxiety.
Preliminary data on treatment response- National Institute on Drug Abuse (NIDA) Quick Screen/Modified ASSIST | pre intervention(after the informed consent), post intervention (at the end of intervention average 8 weeks after the intervention starts), 2 months post-intervention
  The NIDA Quick Screen/Modified ASSIST was designed under the National Institute on Drug Abuse (NIDA)'s Screening for Drug Use in General Medical Settings Resource Guide. The NIDA Quick Screen asks "In the past year, how often have you used the following?" and then lists the frequency of alcohol use, tobacco products, prescription drugs for nonmedical reasons, and illegal drugs. If a woman answered "no" for all drugs in the quick screen, the participant will still be eligible to participate in the study since this study will look into the trajectory of changes of risks over time. If a participant answered "yes" to use of illegal and prescription drugs for nonmedical reasons, the survey proceeded to the NIDA Modified ASSIST, which asked for more detailed use of substances. The range of risk is 0-27+, where 0-3 indicates lower risk, 4-26 indicates moderate risk, and a score ≥27 indicates high risk and the need for referral.